CLINICAL TRIAL: NCT01885052
Title: NCI Young Adult Smoking Cessation Evaluation
Brief Title: Evaluation of National Cancer Institute Young Adult Stop-Smoking Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 999913156; 13-C-N156
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2016-04-27

CONDITIONS: Smoking; Smoking Cessation; Cigarette Smoking; Tobacco, Smoking
Keywords: Smoking Cessation Clinical Trial; Text Messaging Program; Smoking Cessation Aid
MeSH Terms: conditions — Smoking; Smoking Cessation; Cigarette Smoking

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- 1 (Placebo Comparator): Receives weekly assessment messages ONLY
  Interventions: Behavioral: Low Contact
- 2 (Active Comparator): Receives two week countdown messaging to quit date, and weekly assessment messages post quit date
  Interventions: Behavioral: QuitTXT Study
- 3 (Active Comparator): Receives two week countdown messages to quit date, receives mulitiple messages per day post quit date with tips, encouragement and supportive messaging
  Interventions: Behavioral: QuitTXT Study

INTERVENTIONS:
Behavioral: QuitTXT Study — Assess the efficacy of a 6-8 week text message program to help young adults quit smoking.
  Arms: 2; 3
Behavioral: Low Contact
  Arms: 1

SUMMARY:
Background:

- Researchers want to see how well the QuitTXT text-message program helps smokers ages 18 29 stop smoking. This is part of a larger online stop-smoking program by the National Cancer Institute. The QuitTXT program is a 2-week countdown to the smoker s quit date with 6 weeks of follow-up messages. Program participants will receive texts on their cell phones, including tips, information, and motivational messages, and then fill out surveys.

Objectives:

- To study how well the QuitTXT program helps smokers ages 18 29 stop smoking.

Eligibility:

- Adults ages 18 29 who have smoked on at least 5 of the past 30 days and who want to stop smoking in the next 30 days.

Design:

* Participants will receive a certain number of text messages during the 8-week study. They will receive between 0 to 5 messages per day (or up to a total of 130 messages).
* Participants will first fill out a survey about their smoking and quitting experiences. Then they will choose a date to quit smoking (a quit date ) between 2 and 3 weeks after this survey.
* Participants will take four other surveys online, one during the program and three more after they ve completed the program. Each survey will take about 10 20 minutes and asks about their smoking habits and views on smoking and quitting. Each survey will be sent by email, with reminders sent by email or telephone.
* Participants will receive an iTunes or Amazon gift card for completing each survey honestly.

DETAILED DESCRIPTION:
This study seeks to assess the effectiveness of the QuitTXT program, a text message cessation intervention designed for young adult smokers ages 18-29. The QuitTXT program is a component of a larger web-based tobacco cessation intervention resource provided by the National Cancer Institute. The program focuses on providing actionable strategies and fact based information, serving as an engagement tool delivering two-way communication, and delivering intra- and extra-treatment support. The structure of the QuitTXT program is designed as a 14-day countdown to quit date with subsequent six weeks of messages. Throughout the program, users will receive texts that cover a variety of content areas including tips, informational content, motivational messaging, and keyword responses.

The study seeks to recruit a large sample of young adult smokers ages 18-29 to examine how exposure to the QuitTXT program affects participants.

There will be 3-arms to the study:

Participants in Arm 1, the control group of the study, will only receive the weekly assessments asking them of their smoking status.

Participants in Arm 2 will receive a texting program that consists of up to two weeks of countdown to quit messaging plus assessments messages that all groups receive for a total of 8 weeks.

Participants in Arm 3 will receive the full text messaging program.

All groups will be able to select a quit date within a 7-day window (between 2 and 3 weeks after they complete the baseline survey). Participants in Arm 3 will receive motivational/informational messages while participants in group 1 will receive only assessment messages. Participants in Arm 2 will receive the countdown messages to their quit date, but not the motivational messaging after their quit date. Like Arm 1, they will only receive assessment messages after their quit date.

This study will add unique value to the existing literature by teasing out the effect of some messages vs. frequent, motivational/informational messaging on quit rates and intent to quit among young adults.

ELIGIBILITY:
* For this study, we will recruit smokers aged 18 to 29 who have smoked on at least 5 of the last 30 days and who are interested in stopping smoking in the next 30 days. To be eligible, a young adult must meet the following criteria:

Ages 18-29 years

Reside in the US

Smoke cigarettes at least 5 days/month

Be interested in quitting cigarette use

Not be involved in a cessation program

Have an active email account

Be able to receive text messages on their cell phone

Be the only member of your household participating in this study

Be willing to share contact information with the study team in order to share information about the study on a timely basis.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4432 (Actual)
Dates: Start 2013-06-12; Primary Completion 2014-10-12 (Actual); Study Completion 2015-05-28 (Actual)

PRIMARY OUTCOMES:
Quit smoking status | 1, 3, and 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Erik M Augustson, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Armstrong AW, Watson AJ, Makredes M, Frangos JE, Kimball AB, Kvedar JC. Text-message reminders to improve sunscreen use: a randomized, controlled trial using electronic monitoring. Arch Dermatol. 2009 Nov;145(11):1230-6. doi: 10.1001/archdermatol.2009.269. PMID 19917951
- [Background] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Background] Baer JS, Lichtenstein E. Classification and prediction of smoking relapse episodes: an exploration of individual differences. J Consult Clin Psychol. 1988 Feb;56(1):104-10. doi: 10.1037//0022-006x.56.1.104. No abstract available. PMID 3346434
- [Derived] Squiers L, Brown D, Parvanta S, Dolina S, Kelly B, Dever J, Southwell BG, Sanders A, Augustson E. The SmokefreeTXT (SFTXT) Study: Web and Mobile Data Collection to Evaluate Smoking Cessation for Young Adults. JMIR Res Protoc. 2016 Jun 27;5(2):e134. doi: 10.2196/resprot.5653. PMID 27349898